CLINICAL TRIAL: NCT01613313
Title: A Dose Escalation Study Using Collagenase Clostridium Histolyticum in the Treatment of Lipoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zachary Gerut (Individual)
Collaborators: Advance Biofactures Corporation (Industry)
Responsible Party: Sponsor-Investigator, Zachary Gerut, Sponsor-Investigator, Gerut, Zachary, M.D.
Organization: Gerut, Zachary, M.D. (Individual)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lipoma DE/01
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Lipoma
Keywords: Lipoma; Fatty Tumor
MeSH Terms: conditions — Lipoma | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose #1 (Experimental): single injection 0.058 mg Collagenase Clostridium Histolyticum
  Interventions: Drug: Collagenase Clostridium Histolyticum
- Dose #2 (Experimental): single injection 0.15 mg Collagenase Clostridium Histolyticum
  Interventions: Drug: Collagenase Clostridium Histolyticum
- Dose #3 (Experimental): single injection 0.29 mg Collagenase Clostridium Histolyticum
  Interventions: Drug: Collagenase Clostridium Histolyticum
- Dose #4 (Experimental): single injection 0.44 mg Collagenase Clostridium Histolyticum
  Interventions: Drug: Collagenase Clostridium Histolyticum

INTERVENTIONS:
Drug: Collagenase Clostridium Histolyticum — This is a dose escalation study in which subjects will sequentially receive single injections of 0.058 mg, 0.15 mg, 0.29 mg, 0.44 mg.
  Other Names: XIAFLEX

SUMMARY:
The purpose of this research is to evaluate the safest and most effective dose of a Food and Drug Administration (FDA) approved drug (XIAFLEX) in the treatment of lipoma (fatty tumors of varying sizes that occur commonly in the adult population). The fat in the lipoma is like normal fat except that it is enclosed in a balloon-like structure which is made of collagen (fibrous tissue). Treatment of the lipoma with an injection of XIAFLEX (a protein that breaks down collagen fibers) may dissolve the collagen/fibrous strands thereby decreasing the size of the lipoma or removing it.

DETAILED DESCRIPTION:
Lipomas are common mesenchymal, benign, fatty tumors of varying sizes that occur in the general adult population. They usually present as painful or annoying lumps that are palpable and often visible in the subcutaneous tissue. Many subcutaneous lipomas are asymptomatic and are removed for non-medical reasons. However, they may cause the subject pain or discomfort or interfere with normal activity.

Spontaneous remission of lipomas has not been reported. A lipoma, once it presents itself, remains there for the lifetime of a person who carries it and may stay small or become larger. Alternative treatments of the lipoma are surgery or liposuction. If a large excision is performed there is the problem of having a very large scar and the accompanying issues of healing a large scar, or possible formation of a hematoma followed by consolidation of the hematoma and the remnants of a mass of scar tissue. This is often painful and more problematic than the original lipoma. liposuction also has the potential for hematoma formation followed by scar mass residual.

To avoid the complications listed above, a non-invasive method of treatment, such as enzyme mediated disassociation of adipose tissue, would be desirable. The primary aim of this study is to perform a step-wise approach in dosing to evaluate the safety and efficacy of clostridium histolyticum as a non-operative treatment for lipoma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history lipoma at least one year and no treatment within last 90 days
* Lipoma diagnosed as benign
* Lipoma is a single mass with easily definable edges
* Lipoma has an area of 2.0 to 17 cm squared
* Women of childbearing potential must use an acceptable method of birth control

Exclusion Criteria:

* Lipomas on the head, neck, hand or foot, or female breast
* Women who are nursing or pregnant
* Subjects who have participated in any investigational drug trial within 45 days of enrollment in this study
* Subjects with known allergy to collagenase or any of the inactive ingredients in XIAFLEX
* Subjects with diabetes or any medical condition that would make the subject unsuitable for enrollment.
* Subjects having a history of trauma in the area of the lipoma
* Subjects with a history of connective tissue diseases or rheumatological diseases.
* Subjects with uncontrolled hypertension
* Subjects currently receiving or planning to receive anticoagulant medication except for less than 150 mg aspirin daily and over-the-counter nonsteroidal anti-inflammatory drugs) within 7 days before injection of study drug
* Subjects having the following laboratory abnormalities:
* ALT/AST greater than 3 times the upper limit of normal
* Creatinine greater than 2
* Hemoglobin/hematocrit and WBC outside the normal range

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary E Gerut, M.D., Principal Investigator — Gerut, Zachary, M.D.
Locations (1):
- Zachary E. Gerut, M.D., Hewlett, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 1 site in the United States
Period: Overall Study
Arm/Group | Dose #1 | Dose #2 | Dose #3 | Dose #4
Started | 2 | 4 | 4 | 4
Completed | 2 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose #1 | Dose #2 | Dose #3 | Dose #4 | Total
Number analyzed (Participants) | 2 | 4 | 4 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.0 (5.66) | 51.5 (12.50) | 41.3 (11.09) | 57.0 (4.97) | 49.6 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 1 | 9
  Male | 0 | 1 | 1 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 4 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Visible Surface Area of the Lipoma
Description: The primary efficacy outcome is the visible surface area of the lipoma measured as the longest dimension (length) times the longest dimension perpendicular to length (width). Visible surface area will be determined by caliper and will be analyzed as the percent change from baseline at the 6-month post injection visit.
Time Frame: Baseline and Six months post injection of study drug
Population: Analysis population consists of all subjects who were enrolled and received the administration of study drug.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Dose #1 | Dose #2 | Dose #3 | Dose #4
Number analyzed (Participants) | 2 | 4 | 4 | 4
Percent change from baseline | -31.69 (80.83) | -47.57 (23.48) | -52.42 (50.61) | -66.60 (17.82)
Statistical Analysis 1: Comparison: Dose #1 vs Dose #2 vs Dose #3 vs Dose #4; This is a proof of concept dose escalation study. No power justification has been implemented. Descriptive data provided for each arm; Test type: Superiority or Other; No p value; Mean Difference (Final Values) = 50

2. Secondary Outcome: Relative Change in Volume of the Lipoma
Description: A secondary outcome is the relative change in volume of the lipoma as determined by MRI. This outcome will be analyzed as the change from baseline to 6 months post injection.
Time Frame: Baseline and 6 months post injection of study drug
Population: Analysis is based on the population that consists of all subjects who are enrolled and received administration of study drug
Measure: Mean (Standard Deviation); unit: Percent reduction from baseline
Arm/Group | Dose #1 | Dose #2 | Dose #3 | Dose #4
Number analyzed (Participants) | 2 | 4 | 4 | 3
Percent reduction from baseline | -54.16 (34.3) | -62.33 (30.39) | -11.35 (32.12) | -34.75 (24.21)
Statistical Analysis 1: Comparison: Dose #1 vs Dose #2 vs Dose #3 vs Dose #4; This is a proof of concept dose escalation study. No power of justification was implemented. Descriptive statistics was provided for each arm only; Test type: Superiority or Other; Mean Difference (Final Values) = 50

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Day 0 through 6 months post administration of study medication
Arm/Group | Dose #1 | Dose #2 | Dose #3 | Dose #4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/2 | 3/4 | 3/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose #1 (N=2) | Dose #2 (N=4) | Dose #3 (N=4) | Dose #4 (N=4)
Bruising (General disorders) | 1 | 3 | 3 | 4 — Injection site reaction
Pain (General disorders) | 0 | 3 | 1 | 3 — Injection Site
Swelling (General disorders) | 0 | 0 | 3 | 1 — Injection site
Contusion (Vascular disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dizziness (Cardiac disorders) | 0 | 0 | 1 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other